CLINICAL TRIAL: NCT04651868
Title: The Effect of Exogenous Glucagon-like Peptide 2 on Cholecystokinin-induced Gallbladder Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-20039104
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Gallbladder
Keywords: Glucagon-Like Peptide 2; Gallbladder; Gallbladder Motility

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Day A, B, C and D will be conducted in a randomized and double-blinded order (blinded for the participant and the investigator). The infusion order will be unblinded after the last patient last visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CCK + GLP-2 (Experimental): A 180 mins intravenous infusion with cholecystokinin (0.4 pmol × kg^-1 × min^-1) and a 210 mins intravenous infusion with GLP-2 (10 pmol × kg^-1 × min^-1)
  Interventions: Other: GLP-2; Other: CCK
- CCK + placebo (Experimental): A 180 mins intravenous infusion with cholecystokinin (0.4 pmol × kg^-1 × min^-1) and a 210 mins intravenous infusion with isotonic NaCl
  Interventions: Other: Placebo; Other: CCK
- Placebo + GLP-2 (Experimental): A 180 mins intravenous infusion with isotonic NaCl and a 210 mins intravenous infusion with GLP-2 (10 pmol × kg^-1 × min^-1)
  Interventions: Other: GLP-2; Other: Placebo
- Placebo + placebo (Experimental): A 180 mins intravenous infusion with isotonic NaCl and a 210 mins intravenous infusion with isotonic NaCl
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLP-2 — A 210 mins intravenous infusion with GLP-2 (10 pmol × kg^-1 × min^-1)
  Arms: CCK + GLP-2; Placebo + GLP-2
Other: Placebo — A 210 mins intravenous infusion with isotonic NaCl
  Arms: CCK + placebo; Placebo + placebo
Other: CCK — A 180 mins intravenous infusion with cholecystokinin (0.4 pmol × kg^-1 × min^-1)
  Arms: CCK + GLP-2; CCK + placebo
Other: Placebo — A 180 mins intravenous infusion with isotonic NaCl
  Arms: Placebo + GLP-2; Placebo + placebo

SUMMARY:
The study is a randomized, double-blinded, placebo-controlled, cross-over study, which will investigate the acute effects of the gut-derived hormone glucagon-like peptide 2 (GLP-2) on cholecystokinin (CCK)-induced gallbladder emptying. Furthermore, the investigators will investigate different hormonal responses and appetite during the study days.

The investigators hypothesize that GLP-2 will overrule the potent gallbladder relaxing effect of CCK.

We will include 15 healthy male participants, and each of the participants will participate in four study days. GLP-2 and CCK will be given intravenously, and will be placebo-controlled. Gallbladder volume will be determined by frequent ultrasonography scans. Appetite will be assessed by Visual Analog Scales through out the study day and an ad libitum meal at the end of the study day. Blood samples will be drawn at regular intervals to asses different hormonal responses.

DETAILED DESCRIPTION:
Background

AIM OF THE STUDY The aim of the study is to investigate if exogenous GLP-2 can overrule CCK-induced gallbladder contraction

STUDY DESIGN The study is a randomized, double-blinded, placebo-controlled, crossover study enrolling 15 healthy participants. Each participant will undergo four separate study days in randomized order. Each study day encompasses two intravenous (iv) infusions, one with CCK (0.4 pmol × kg^-1 × min^-1) or placebo (saline), and one with GLP-2 (10 pmol × kg^-1 × min^-1) or placebo (saline): Day A, CCK + GLP-2; Day B, CCK + placebo; Day C, placebo + GLP-2; Day D, placebo + placebo.

METHODS For each participant, the study consists of an information visit, a screening visit and four experimental days within a time period of minimum 2 months, and with a minimum of three days between each experimental day with procedures explained below.

RECRUITMENT OF PARTICIPANTS Relevant persons, who have previously participated in trials at the investigators research facility and at that time accepted to be contacted again regarding other research projects will be contacted by telephone or e-mail. Alternatively, advertisements regarding the project will be published at www.forsoegsperson.dk, other relevant internet / social media pages and/or local or national newspapers. Persons responding positively will receive the written information. A couple of days after receiving the written information, the potential participant will be contacted and, if the person is still interested in participating, an information visit will be arranged. If the person decides to participate, written consent will be obtained. Obtaining of written consent will be postponed if the potential participant requires more time for consideration. After obtaining written consent the date for the screening visit is planned.

EXPERIMENTAL DAYS All experiments are carried out at the investigators research facility at Center for Clinical Metabolic Research at Gentofte Hospital, where all the necessary equipment and expertise are available. If participants have any ongoing medical treatment, the participant will be informed to pause the treatment one week prior to each experimental day. The duration of each experimental day will be approximately 5 hours.

After arriving at the research facility after an overnight (10h) fast (including water, coffee and medicine), the participant will be asked to empty the urinary bladder and two urine samples are collected. Two intravenous (iv) catheters will then be inserted in the cubital veins (one in each arm). One for collection of blood samples and one for administration of CCK/placebo and GLP-2/placebo. The forearm from which blood samples are drawn will be wrapped in a heating pad (40-45°C) throughout the experiment for arterialisation of venous blood. The participant will rest approximately 30 minutes before start of the experimental procedures. At time 0 min, CCK/placebo infusion will be started. At time 30 min, the GLP-2/placebo infusion will be started. At time -15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 195, 210 and 240 min, gallbladder height, width and length will be determined by ultrasonography scans for evaluation of gallbladder volume (calculated by the ellipsoid method). Blood samples will be collected at time -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 min. Blood pressure and heart rate will be measured at time -15, 0, 30, 60, 90, 120, 150, 180 and 240 min. The appetite of the participants will be assessed by Visual Analogue Scale (VAS) at time -15, 0, 15, 45, 75, 105, 135, 180, 210 and 240 min. At time 180 min the CCK/placebo infusion will be stopped. At time 240 min the GLP-2/placebo infusion will be stopped. At 240 min, the participants receive a standardized ad libitum meal consisting of minced meat, pasta, corn, carrots, peppers, cream and salt and pepper. Participants are instructed to eat as much as they can until they feel comfortably full. The meal is to be consumed within 30 minutes, and before and after the appetite of the participants will be evaluated by VAS. After the meal the participant will again be asked to empty the urinary bladder and two urine samples will be collected.

Data from the study days will be recorded in Clinical Report Forms.

LABORATORY METHODS For bedside measurement of plasma glucose, blood will be sampled into sodium-fluoride-coated tubes, centrifuged immediately at room temperature and analysed on a glucose analyzer. For analysis of plasma concentrations of gut-derived hormones degraded by DPP-4 blood will be collected in chilled tubes (on ice) containing EDTA and the specific DPP-4 inhibitor valine-pyrrolidide (0.01 ml of 1 mmol/l valine-pyrrolidide solution - 4.3 mg in 20 ml sterile water/ml blood). For analysis of serum concentrations of other secondary endpoints blood will be sampled in plain tubes with clot activator for coagulation (10 minutes at room temperature). EDTA and plain tubes will be centrifuged for 15 minutes and 4°C. Plasma/serum samples will be stored at -20°C or -80°C until analysis.

STATISTICS AND CALCULATIONS Data will be processed and presented with the use of standard descriptive statistics. Area under the curve (AUC) will be calculated by use of the trapezoid rule. Results will be reported as mean and standard deviation (SD) and as baseline subtracted AUC (bsAUC). Normally distributed data will be compared using one-way repeated measurements analysis of variance. Repeated measurement analysis of variance will be used for statistical analysis of repeated measurements in the same participant. Data that are not normally distributed will be analyzed using non-parametric tests. P values <0.05 will be considered statistically significant, i.e. significance level (α) of 5%. Power of the study (1-β) is set to 80%, where β (20%) is the risk of accepting a hypothesis that is false.

The population size (N) has been calculated using the formula:

N = (Za + Zb)^2 × (SD^2)/(MIREDIF^2), where Za is a table value according to a two-sided standard normal distribution (1.96), Zb is a table value according to a one-sided standard normal distribution (0.84). MIREDIF is the minimum relevant difference. SD and MIREDIF are assessed as bsAUC for gallbladder volume.

The investigators plan to enroll 15 participants. In a previous study with CCK-induced gallbladder emptying bsAUC (0-120) for gallbladder volume was -1791 ml × min and SD 795.2 ml × min. Based on these values a 30 % difference in bsAUC for gallbladder volume can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Male gender
* Age 18-65 years
* Body mass index (BMI) 18.5-24.9 kg/m2
* Fasting plasma glucose ≤6 mmol/l and glycated haemoglobin (HbA1c) ≤ 42 mmol/mol
* Normal hemoglobin (males 8.3-10.5 mmol/l)
* Informed and written consent

Exclusion Criteria:

* Nephropathy (eGFR < 90 ml/min/1.73m2 and/or albuminuria)
* Known liver disease and/or alanine aminotransaminase (ALAT) and/or aspartate transaminase (ASAT) > 2 × upper normal reference limit
* Active or recent (within 5 years) malignant disease
* Any history of colon cancer
* Treatment with medicine that cannot be paused for 1 week
* Active tobacco smoking
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Gallbladder volume | 0 to 240 minutes
  Baseline subtracted area under the curve for gallbladder volume

SECONDARY OUTCOMES:
Maximum gallbladder ejection fraction | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 195, 210 and 240 minutes
  Calculated on the basis of gallbladder volume time curves.
GLP-2 | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of GLP-2
CCK | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of CCK
Bile Acids | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of bile acis
Cholesterols | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of cholesterols
Triglycerides | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of triglycerides
Insulin | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of insulin
C-peptide | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Plasma measurement of C-peptide
Plasma glucose | -15, 0, 10, 30, 40, 50, 70, 100, 140, 180, 210 and 240 minutes
  Measurement of plasma glucose
Appetite | -15, 0, 15, 45, 75, 105, 135, 180, 210 and 240 minutes
  Answers to Visual Analog Scales regarding hunger, satiety etc.
Appetite | 240-270 minutes
  Meal ingestion (gram)
Blood pressure | -15, 0, 30, 60, 90, 120, 150, 180 and 240 minutes
  Non invasive blood pressure measurement
Heart rate | -15, 0, 30, 60, 90, 120, 150, 180 and 240 minutes
  Non invasive heart rate measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nina L Hansen, MD, Principal Investigator — Center for Clinical Metabolic Research, Genofte University Hospital
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lange AH, Hansen NL, Pedersen MG, Nerild HH, Rehfeld JF, Hartmann B, Holst JJ, Ellegaard AM, Knop FK. Exogenous Glucagon-like Peptide 2 Counteracts Exogenous Cholecystokinin-induced Gallbladder Contraction in Healthy Men. J Clin Endocrinol Metab. 2024 Dec 18;110(1):123-129. doi: 10.1210/clinem/dgae421. PMID 38888179